CLINICAL TRIAL: NCT05846620
Title: Pulmonary Immune Cell-microbiome Interactions in the Healthy Lung: the ILLUMINA-2 Study
Brief Title: Pulmonary Immune Cell-microbiome Interactions in the Healthy Lung
Acronym: ILLUMINA-2
Status: Recruiting | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ronni R. Plovsing, Associate professor, Senior Consultant of ICU, Hvidovre University Hospital
Other Study IDs: H-22046545
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: healthy lung, lung microbiota, microbiome
MeSH Terms: interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, BAL fluid, endotracheal aspirate, oral/nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women
  Interventions: Procedure: Bronchoalveolar lavage
- Men
  Interventions: Procedure: Bronchoalveolar lavage

INTERVENTIONS:
Procedure: Bronchoalveolar lavage — Bronchoalveolar lavage in the middle lobe of the right lung and a mini-bronchoalveolar lavage in the upper and lower lobe of the right lung

SUMMARY:
The overall aim is to to provide a normal material for the composition and spatial heterogeneity of the following in the healthy lung: i) immune cell populations and their activation patterns, ii) the surrounding cytokine-chemokine milieu, including trans-compartmental fluxes of these mediators between the lung and bloodstream, and iii) the lung microbiome.

Main hypotheses:

* Absolute and relative immune cell counts in bronchoalveolar lavage fluid (BALF) are similar to those previously reported by other methods6,7.
* No trans-compartmental flux of cytokines between the lungs and bloodstream is present, but cytokine concentrations (notably IL-6 and IL-8) vary with the immune-cell-microbiome composition.
* Immune cell (mainly T cell) activation, differentiation, and gene expression patterns are expected to differ between blood and BALF in a manner that depends on the regional diversity of the pulmonary microbiome.

DETAILED DESCRIPTION:
The coronavirus disease 2019 pandemic, caused by severe acute respiratory syndrome coronavirus 2, has brought with it several studies on the local pulmonary immune system, which was until very recently largely a terra incognita. With these new methods, apparently fundamental aspects of lung disease have been uncovered, including pulmonary hyper inflammation. However, very little is currently known about the composition of the normal immune cell population in the human lung, including its interplay with the pulmonary microbiome, that is, the commensal microbiota of interacting bacteria and fungi that reside within the healthy lung

Overall design: In 50 patients (25 males, 25 females), intubated for elective surgery in general anaesthesia, an endotracheal aspirate and BAL fluid (BALF) from separate lung segments will be obtained. Furthermore, an oral and nasal swab and blood samples will be collected. This will be done immediately after intubation.

The following is obtained from the patient's electronic health record: diagnosis codes and medication (type and dosage), smoking history (current/previous/never smoker; pack years), type of operation; furthermore, the health record is screened for any exclusion criteria

Blood samples are drawn from the patient's peripheral venous catheter (inserted for clinical purposes) immediately before BALF collection.

Bronchoscopy with BALF collection: This procedure is performed in a standardized fashion according to current clinical guidelines. Immediately prior to the procedure, an oral swab, nasal swab and an endotracheal aspirate (ETA) are obtained. FIO2 is then increased to 1.0, and the bronchoscopy procedure is performed using a disposable videoscope with an outer diameter of 5.0 mm). Three successive 50-ml aliquots of prewarmed (37°C) isotonic saline are instilled in the medial segment of the right middle lobe, aspirated immediately with low negative suction pressure (< 100 cm H2O), and pooled into a sterile glass container on ice to obtain a BALF specimen.

Afterwards a mini-BAL is performed in the upper and lower lobe of the right lung with a single installation of 20 ml isotonic saline in each lobe with immediately aspiration into a sterile container.

Measurements: The composition of the immune cell population, as well as the function and differentiation of various cell lines will be investigated by single-cell RNA sequencing (scRNA-seq) on selected immune cells from BALF, ETA, and blood, and this will be supplemented by bulk RNA sequencing with sample barcoding and multiplexing, giving a detailed expression pattern of all samples.

The composition microbiome in BALF, ETA, and oral swabs will be assessed by targeted amplicon sequencing of the hyper-variable regions 1 through 3 of the 16S subunit of ribosomal RNA gene for bacteria.

Statistical analyses: will be performed using R statistical software version 4.1.1 (R Project for Statistical Computing) within RStudio statistical software version 1.4.1717 (RStudio), and p<0.05 considered statistically significant. Inspection of normality and variance homogeneity will be done by creating qq-plots and histograms. The statistical inference tools SPIEC-EASI and HeatMaps will be used, and based on correlational analyses, principal component analyses, including non-hierarchal cluster analysis, will be applied to identify traits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 40 to 75

Exclusion Criteria:

* Immune deficiency
* Lung disease
* Active cancer or infection
* Absolute contraindications for bronchoscopy

  * Untreated malignant arrhythmia
  * Documented or suspected intracranial hypertension (intracranial pressure ≥ > 15 mmHg)
  * One-lung ventilation
  * Severe coagulopathy

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients referred for elective surgery requiring intubation at Hvidovre Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Lung microbiome | Day 0 (subsequent to study inclusion)
  16S ribosomal RNA (rRNA) and 18S rRNA PCR for bacterial or fungal pathogen identification in bronchoalveolar lavage fluid
Lymphocyte populations | Day 0 (subsequent to study inclusion)
  Cell populations and subpopulations evaluated by 10 colored flow cytometry (B cells, T cells, TCR subsets, Tregs/Th17, dendritic cells, myeloid cells and neutrophils) in bronchoalveolar lavage fluid and blood

SECONDARY OUTCOMES:
Cell differential counts and cytomorphological analyses of BALF | Day 0 (subsequent to study inclusion)
Trans-compartmental fluxes | Day 0 (subsequent to study inclusion)
  (calculated from plasma- and urea-adjusted BAL)
Auto-antibodies against tI-IFNs in blood | Day 0 (subsequent to study inclusion)
  Measured in bronchoalveolar lavage fluid
White blood cells counts | Day 0 (subsequent to study inclusion)
  Total white blood cells, neutrocytes, lymphocytes, and monocytes in bronchoalveolar lavage fluid and blood
Cytokines | Day 0 (subsequent to study inclusion)
  Multiplex assay for measuring cytokines in bronchoalveolar lavage fluid and plasma (e.g. IL-1-beta, IL-1RA, IL-2, IL-6, IL-8, IL-10, IL-17, IL-18, IL-33, IL-35, TGF-beta, TNF-alpha, HMGB1)
Number and characterizations of respiratory pathogens | Day 0 (subsequent to study inclusion)
  Respiratory film array PCR for testing for number of pathogens
Number and characterizations of microorganisms | Up to 12 weeks
  Growth of pathogenic microorganisms in body fluids (e.g. urine, blood, bronchoalveolar lavage fluid) in microbiological assays

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Berg, MD PhD, Study Chair — Biomedical Science of Health, University of Copenhagen
Locations (1):
- Hvidovre Hospital, University of Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided